CLINICAL TRIAL: NCT05148390
Title: Prospective Observational Explorative Study to Examine Clinical Performance and Safety of Cutimed® Gelling Fiber in Routine Clinical Practice
Brief Title: Study to Examine Clinical Performance and Safety of Cutimed® Gelling Fiber in Routine Clinical Practice
Acronym: GELFI
Status: Completed | Type: Observational
Sponsor: BSN Medical GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: C2820
Record Dates: First submitted 2021-11-05; First posted 2021-12-08 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2023-11

CONDITIONS: Leg Ulcer; Diabetic Foot Ulcer; Pressure Ulcer; Surgical Wound; Abrasion; Laceration; Burn, Partial Thickness; Oncology Wound
MeSH Terms: conditions — Leg Ulcer; Diabetic Foot; Pressure Ulcer; Surgical Wound; Lacerations; Burns

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Cutimed® Gelling Fiber — application of dressing

SUMMARY:
This is a post - market study with a wound dressing, a CE-marked medical device available on the european market. The device will be used in routine clinical practice, i.e. within its intended purpose and without any additional invasive or stressing examinations for the patients.

Up to 36 adult patients with wounds suitable to be treated with the medical device and meeting the inclusion/exclusion criteria will be enrolled at two participating German sites.

During 5 on-site visits within 28 days routine weekly dressing changes the Health Care Professional will examine the wound and will perform required wound care and dressing changes. Pictures of the wound with and without dressing will be taken at each visit and used for automatic analysis. The subjects will be asked to rate their general wound pain and the pain perceived during dressing changes. A wound-related quality of life questionnaire will be presented to the subjects twice and the subject and HCP will rate their safisfaction with the product.

DETAILED DESCRIPTION:
This Post Market Clinical Follow up (PMCF) study will examine product features of the CE-marked wound dressing after having received market authorization regarding the fulfilment of predefined requirements for the successful management of skin integrity during wound care. The primary purpose of this study is to evaluate clinical safety and performance of the product when used on several wounds in routine wound care without any additional invasive or burdensome methods and within the intended use.

As primary objective the dressing´s absorption performance and its ability to prevent exudate accumulation in the wound will be investigated. Further, device disintegration, need of debridement, wound and skin conditions, treatment related pain, general wound pain, dressing adhesion and quality of life as well as Helath Care professional's (HCP´s) and patient´s satisfaction are considered as secondary outcomes.

In total, 36 eligible subjects will be enrolled at 2 German sites, including 15 % dropouts.

5 on-site visits are to be performed by the subjects in the scope of routine weekly wound care/dressing change visits during 28 days (Day 0, Day7, Day 14, Day21, Day28). The IMD will be applied during each on-site visit including wound care, wound examination/documentation and dressing change according to HCP's judgment and individual circumstances of the wound. Photographic documentation of the wound and the wound with applied dressings will be performed and used for further automatic wound/tissue analyis. General wound pain as well as pain perceived during dressing change will be documented, as well as Wound-related Quality of life as well as Patient's/HCP's satisfaction with the product.

ELIGIBILITY:
Inclusion Criteria:

* mentally and physically able to participate in study
* written informed consent to participate in the study
* Diagnosed wound indicated for treatment with Cutimed® Gelling Fiber for 4 weeks (except for internal body cavities and closed wounds)
* Subjects with more than one ulcer are eligible for inclusion, however only one ulcer per subject will be included in the study.

Exclusion Criteria:

* Sensitivity to or allergic reaction to the dressing or its components
* Participation in any other clinical study investigating drugs or medical devices
* Subjects presenting with wounds including internal body cavities or closed wounds
* Alcohol and drug addiction
* Pregnant or breast-feeding subjects
* Underlying diseases are not treated according to respective country-specific guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Representativeness of the investigation population is assumed to be high in relation to the target population since this is a PMCF study, where the IMD will be used within the intended purpose including the intended patient population. Therefore, the IMD will be tested by the population for whom it is in fact intended for once placed on the market among other intended users. Inclusion and exclusion criteria are aligned with the product´s intended purpose.
  No vulnerable subjects such as children, pregnant women, or sponsors or manufacturers staff will participate in this study guaranteed by specific inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2022-04-24 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2023-07-26 (Actual)

PRIMARY OUTCOMES:
Exudate absorption by IMD ('yes', 'no') | day 7
  Percentage of subjects with exudate absorbed by the IMD per visit
Exudate absorption by IMD ('yes', 'no') | day 14
  Percentage of subjects with exudate absorbed by the IMD per visit
Exudate absorption by IMD ('yes', 'no') | day 21
  Percentage of subjects with exudate absorbed by the IMD per visit
Exudate absorption by IMD ('yes', 'no') | day 28
  Percentage of subjects with exudate absorbed by the IMD per visit
Exudate accumulation in the wound by IMD ( 'no', 'minimal amount', 'medium amount', 'high amount') | day 7
  Percentage of subjects with remaining exudate in wound per amount and visit
Exudate accumulation in the wound by IMD ( 'no', 'minimal amount', 'medium amount', 'high amount') | day 14
  Percentage of subjects with remaining exudate in wound per amount and visit
Exudate accumulation in the wound by IMD ( 'no', 'minimal amount', 'medium amount', 'high amount') | day 21
  Percentage of subjects with remaining exudate in wound per amount and visit
Exudate accumulation in the wound by IMD ( 'no', 'minimal amount', 'medium amount', 'high amount') | day 28
  Percentage of subjects with remaining exudate in wound per amount and visit

SECONDARY OUTCOMES:
Changes in need for debridement | Throughout days 0, 7, 14, 21 and 28
  Percentage of subjects with need for debridement per visit
Changes in debridement ease | Throughout days 0, 7, 14, 21 and 28
  Percentage of subjects per debridement ease ('easy', 'moderate', 'heavy', 'not applicable') per visit
Changes in wound margin condition | Throughout days 0, 7, 14, 21 and 28
  Percentage of subjects per wound margin condition('intact', 'macerated', 'redness', 'ragged') per visit
Changes in peri-wound skin condition | Throughout days 0, 7, 14, 21 and 28
  Percentage of subjects per peri-wound skin condition ('intact', 'macerated', 'redness', 'dry/flaky', 'edematous' ,'weeping') per visit
Changes in wound tissue type | Throughout days 0, 7, 14, 21 and 28
  Percentage of subjects per wound tissue type ('epithelialization tissue', 'granulation tissue', 'slough', 'eschar/necrotic tissue', 'other') per visit
Ease of application | Throughout days 0, 7, 14, 21 and 28
  Percentage of subjects per ease of application ('very easy', 'easy', 'difficult', 'very difficult') per visit
Conformability during application | Throughout days 0, 7, 14, 21 and 28
  Percentage of subjects per conformability ('very good', 'good', 'poor', 'very poor') per visit
Ease of removal | Throughout days 7, 14, 21 and 28
  Percentage of subjects per ease of removal ('very easy', 'easy', 'difficult', 'very difficult') per visit
Dressing adherence on removal | Throughout days 7, 14, 21 and 28
  Percentage of subjects per adherence ('none', 'minor', 'moderate', 'marked') per visit
Pain on removal | Throughout days 7, 14, 21 and 28
  Mean pain perceived by subject using a pain ruler (scale 0-10) per visit
Changes in wound-pain | Throughout days 7, 14, 21 and 28
  Mean pain perceived by subject using a pain ruler (scale 0-10) per visit
Changes in Wound-quality of life Wound-QoL | Day 0 and Day 28
  percentage change in Wound-QoL total scores and subscale scores ('body', 'psyche', 'everyday life' and standalone item) between both visits
HCP Overall satisfaction | day 28
  Percentage per HCP overall satisfaction category ('Very good', 'Good', 'Satisfactory', 'Sufficient', 'Insufficient') for final visit
Subject Overall satisfaction | day 28
  Percent of patient overall satisfaction category ('Very good', 'Good', 'Satisfactory', 'Sufficient', 'Insufficient') for all patients at visit 5
Incidence of adverse events related to IMD | Throughout days 0, 7, 14, 21 and 28
  Total occurence of IMD related adverse events
Incidence of device disintegration (removability in one piece) | Throughout days 0, 7, 14, 21 and 28
  Total occurence of IMD disintegration during removal

CONTACTS AND LOCATIONS:
Overall Officials: Arne Böhling, Dr., Study Director — BSN Medical GmbH
Locations (1):
- Christliches Klinikum Melle GmbH, Unfallchirurgie, Melle, Germany

IPD SHARING:
Plan to Share IPD: No